CLINICAL TRIAL: NCT04674995
Title: Stent Versus Balloon Dilatation in Patients With Tracheal Benign Stenosis
Acronym: STROBE
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio18
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Tracheal Stenosis
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stent: Patients with tracheal stenosis treated with stent placement via rigid bronchoscopy.
  Interventions: Procedure: Stent placement
- Balloon dilatation: Patients with tracheal stenosis treated with balloon dilatation via laryngoscope.

INTERVENTIONS:
Procedure: Stent placement — All interventional procedures have been performed in the operating room with a Dumon rigid bronchoscope under general anesthesia. Neodymium-doped yttrium aluminium garnet laser photoresection was performed at 15-30 watts and pulse duration of 0.5-1.0s whenever indicated. A silicone stent was placed.
  Groups: Stent

SUMMARY:
This is a retrospective, observational cohort study carried out in two operative Units of the University Hospital of Modena (Italy): the Diagnostic and Interventional Bronchoscopy Unit (Unit A) and the Otolaryngology Unit (Unit B). The two units have different protocols routinely applied to treat tracheal benign stenosis. In Unit A, endoscopic treatment is performed through mechanical dilatation via rigid bronchoscopy and further stent placing while in Unit B the endoscopic treatment is performed through balloon dilatation via direct laryngoscopy. The primary purpose was to compare the efficacy of the two technique on tracheal stenosis treatment over time. Patients were defined as "cured" if during the 2 years after 12 months since the last intervention they did not present any of the following: respiratory symptoms, need for a re-intervention or stenosis instability.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* exclusion from resection-anastomosis surgery after multidisciplinary evaluation,
* Cotton Meyer > grade II,
* follow-up of at least 3 years after endoscopic surgery,
* no previous tracheal surgery.

Exclusion Criteria:

* age > 80,
* stent intolerance which requires removal in the first year after endoscopic treatment,
* performance status > 2,
* end-stage chronic pulmonary disease,
* life-threatening stenosis that needs urgent endoscopic treatments,
* any neoplastic stenosis of the airways,
* dynamic etiology of tracheal benign stenosis (excessive dynamic airway collapse, tracheobronchomalacia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We collected clinical, endoscopic and radiological data of patients with benign tracheal stenosis admitted in two operative Units of the University Hospital of Modena (Italy): The Diagnostic and Interventional Bronchoscopy Unit (Unit A) and the Otolaryngology Unit (Unit B) from November 2012 to November 2017
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Re-stenosis rate over time | 36 months
  Patients were defined as cured if during the 2 years after 12 months since the last intervention they did not present any of the following: respiratory symptoms, need for a re-intervention or stenosis instability.